CLINICAL TRIAL: NCT06195696
Title: Illness Perception and Coping in Kidney Transplant Recipients: a Mixed Research Based on Common Sense Model
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wu Jiangxue (Other)
Collaborators: Zunyi Medical College (Other)
Responsible Party: Sponsor-Investigator, Wu Jiangxue, master's degree student, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Other Study IDs: KLL-2023-466
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplantation; Illness Perception and Coping
Keywords: illness perception; common sense model; kidney transplant; mixed research

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: employs questionnaires — The first phase is a quantitative study that employs a questionnaire to investigate the current state of illness perception and the distribution of coping styles in kidney transplant recipients, and to explore the differences in illness perception between positive coping and negative coping patients after kidney transplantation; The second phase involves a descriptive qualitative study that utilizes face-to-face, semi-structured, in-depth interviews to investigate the causes of differences in illness perceptions of different coping styles in kidney transplant recipients who experience idiosyncrasies.
  Other Names: involves a descriptive qualitative study

SUMMARY:
The goal of this observational study is to learn about the current status of illness perception and the distribution of coping styles in kidney transplant recipients. The main question clarifies the current status and experience of illness perception in post-transplant patients with different coping styles, and aims to provide a reference basis for intervention of illness perception in kidney transplant patients, with the aim of improving their current status of illness perception, optimizing their awareness of treatment management and self-care behaviors, and perfecting the modern medical service system. Participants will describe the main tasks participants will be asked to do.

DETAILED DESCRIPTION:
Aims:This study explores the current status of illness perception and the distribution of coping styles in kidney transplant recipients, clarifies the current status and experience of illness perception in post-transplant patients with different coping styles, and aims to provide a reference basis for intervention of illness perception in kidney transplant patients, with the aim of improving their current status of illness perception, optimizing their awareness of treatment management and self-care behaviors, and perfecting the modern medical service system.Methods:This study is based on the Common Sense Model (CSM), which is the most widely used theory for explaining and predicting disease adaptation and patient self-management behaviors.This study utilizes a mixed-methods research design, specifically the interpretive sequence design, consisting of two phases. The first phase is a quantitative study that employs a questionnaire to investigate the current state of illness perception and the distribution of coping styles in kidney transplant recipients, and to explore the differences in illness perception between positive coping and negative coping patients after kidney transplantation; The second phase involves a descriptive qualitative study that utilizes face-to-face, semi-structured, in-depth interviews to investigate the causes of differences in illness perceptions of different coping styles in kidney transplant recipients who experience idiosyncrasies.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18 and 55 who have received a kidney transplant and have been discharged from the hospital for at least 3 months. Patients must have basic communication skills and be willing to participate in the survey voluntarily by signing the informed consent form.

Exclusion Criteria:

(i) Patients with a history of other malignant tumors; (ii) patients who are participating in other clinical trials or related treatments; (iii) patients with other serious physical diseases; and (iv) kidney transplant patients with psychiatric disorders, serious cognitive impairment, or speech defects that prevent them from cooperating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recipients who underwent kidney transplantation at a tertiary hospital in Zunyi between January 01, 2024 and December 2024 were selected for the study using a convenience sampling method.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the current state of illness perception | 2024.01-2024.12
  Using The general information questionnaire to measure
the distribution of coping styles in kidney transplant recipients | 2024.01-2024.12
  Using Simplified Coping Style Questionnaire to measure
the causes of differences in illness perceptions of different coping styles | 2024.01-2024.12
  UsingThe Brief Illness Perception Questionnaire to measure

IPD SHARING:
Plan to Share IPD: Yes